CLINICAL TRIAL: NCT04743609
Title: Ambulatory Respiratory Tract Infection Survey, Burden of Respiratory Syncitial Virus in the Era of Covid-19
Brief Title: RSV Burden in Outpatient Settings
Acronym: Oursyn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A02876-33
Record Dates: First submitted 2021-01-20; First posted 2021-02-08 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: RSV Infection; Children, Only; Outpatient; Bronchiolitis; Otitis Media; Pneumonia
Keywords: RSV; children; bronchiolitis; otitis; pneumonia
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis; Otitis Media; Pneumonia; Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal samples :
  used for rapid antigen test: Sars cov2, influenza and RSV. Also for multiplex RT-PCR (for a subgroup of 500 patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bronchiolitis: - Children under 24 months of age (≤) with First episode of bronchiolitis.
  Aims :
  - For city physicians: Enrrollment of 1000 children with Bronchiolitis not associated with otitis
  - In the hospital (at pediatric emergencies): Enrrollment of 900 children with bronchiolitis
  Interventions: Diagnostic Test: nasopharyngeal samples
- Acute otitis media: Define with Paradise Criteria) or otorrhea
  Enrrollment only for city physicians :
  * 500 children with Otitis not associated with Bronchiolitis
  * 500 children with Otitis associated with Bronchiolitis
  Interventions: Diagnostic Test: nasopharyngeal samples
- Pneumonia: Defined by the presence of opacity of parenchymal condensation and/or pleural effusion on chest X-ray associated with fever.
  Aims:
  - For city physicians: Enrrollment of 100 children with pneumonia
  - In the hospital (pediatric emergencies): Enrollment of 500 children with pneumonia
  Interventions: Diagnostic Test: nasopharyngeal samples

INTERVENTIONS:
Diagnostic Test: nasopharyngeal samples — rapid antigen test for Sars Cov-2, influenza and RSV. multiplex RT-PCR for a subgroup of 500 patients

SUMMARY:
Strengthening outpatient low respiratory tract infection surveillance to document the burden of Respiratory Syncytial Virus (RSV)

DETAILED DESCRIPTION:
The study protocol is designed with three key components: 1. Build on existing PARI outpatient syndromic surveillance by adding laboratory multiplex testing of LRTI samples (RSV, Influenza, SARS-COV-2) 2. Follow all bronchiolitis through the PARI RWE database and document "patient journey" for 5 years after first medical visit 3. Review the electronic PARI data of three previous seasons in order to document the impact of LRTI attributable to RSV in children < 2 years in France prior to enhanced surveillance

ELIGIBILITY:
Inclusion Criteria:

* children under 24 months of age (≤)
* One of the holders of parental authority signed the consent
* Patient affiliated to a social security scheme (Social Security or Universal Medical Coverage)
* First episode of bronchiolitis defined by
* Age ≤24 months
* At least one symptom from group A and one symptom from group B Group A (one or more)
* Fever >38 °C
* Cough
* Otalgia
* Nasal congestion
* Rhinorrhea
* Coryza
* Dysphagia Group B (one or more)
* whistling
* Crackles
* Rales
* Decrease in respiratory noise
* Shortness of breath
* Dyspnea
* OR Acute purulent otitis media (Paradise Criteria) or otorrhea.
* OR Pneumonia defined by the presence of opacity of parenchymal condensation and/or pleural effusion on chest X-ray associated with fever

Exclusion Criteria:

* Age >24 months
* Refusal by one of the parents
* Not affiliated to a social security system

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children under 24 months old with first episode of bronchiolitis or acute otitis media or pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-01-11 (Estimated); Study Completion 2024-01-11 (Estimated)

PRIMARY OUTCOMES:
RSV proven | day of enrrollement
  Percentage of children with proven RSV disease (bronchiolitis, AOM or pneumonia)

SECONDARY OUTCOMES:
Proportion of Respiratory Tract Infections by RSV Status | day of enrrollement
  Percentage of children with Respiratory Tract Infections by RSV Status
Proportion of Respiratory Tract Infections with SARS-CoV-2 | day of enrrollement
  Percentage of children with Respiratory Tract Infections with SARS-CoV-2
Proportion of associated complications by RSV status | day of enrrollement, 15 days and 6 months
  Percentage of children with associated complications by RSV status
Proportion of AOM by RSV status | day of enrrollement
  Percentage of children with AOM by RSV status
Proportion of pneumonia by RSV status | day of enrrollement
  Percentage of children with pneumonia by RSV status
Score of Quality of life | 15 days and 6 months
  Assessed by the quality of life infant scale (from 0-100, so that higher scores indicate better Health-Related Quality of Life)
Caracteristic of tests | day of enrrollement
  Sensitivity, specificity, positive predictive value, negative predictive value positive and negative likelihood ratio of the SARS-Cov2, influenza A/B and RSV rapid antigenic test compared to the reference test by multiplex RT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rybak A, Levy C, Jung C, Bechet S, Batard C, Hassid F, Zouari M, Cahn-Sellem F, Bangert M, Cohen R. Delayed Bronchiolitis Epidemic in French Primary Care Setting Driven by Respiratory Syncytial Virus: Preliminary Data from the Oursyn Study, March 2021. Pediatr Infect Dis J. 2021 Dec 1;40(12):e511-e514. doi: 10.1097/INF.0000000000003270. PMID 34260480
- [Derived] Lenglart L, Levy C, Basmaci R, Levieux K, Kramer R, Mari K, Bechet S, Launay E, Cohen L, Aupiais C, de Pontual L, Rybak A, Lassoued Y, Ouldali N, Cohen R. Nirsevimab effectiveness on paediatric emergency visits for RSV bronchiolitis: a test-negative design study. Eur J Pediatr. 2025 Feb 1;184(2):171. doi: 10.1007/s00431-025-06008-9. PMID 39893316
- See also: Delayed Bronchiolitis Epidemic in French Primary Care Setting Driven by Respiratory Syncytial Virus: Preliminary Data from the Oursyn Study, March 2021 — https://pubmed.ncbi.nlm.nih.gov/34260480/